CLINICAL TRIAL: NCT00160654
Title: A Phase IV, Open-label, Multi-center, Community-based Trial in Asia Studying the Safety and Efficacy of Keppra™ as Adjunctive Therapy in Adult Subjects With Uncontrolled Partial Epilepsy.
Brief Title: Open Label Safety and Efficacy Study of Levetiracetam in Patients With Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01036
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; Partial Onset Seizures; Keppra; Levetiracetam
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levetiracetam (Experimental): Subjects received open-label Levetiracetam.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — * Pharmaceutical form: oral tablets
  * Concentration: 500 mg
  * Route of administration: Oral use
  Other Names: Keppra

SUMMARY:
Community based study assessing safety and efficacy of levetiracetam in partial onset seizures.

The optimal dose in daily clinical practice will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with epilepsy experiencing partial seizures, whether or not secondarily generalized.
* Subjects must present between 3 and 42 partial seizures over the three months prior to protocol Visit 1.
* Use of one (1), but no more than two (2) concomitant marketed antiepileptic drugs (AEDs) at the time of trial entry.

Exclusion Criteria:

* Subjects on vigabatrin, whose visual field has not been assessed as per recommendation of the manufacturer, i.e. every 6 months.
* Presence of known pseudoseizures within the last year.
* Presence of progressive cerebral disease, any other progressively degenerative neurological disease, or any cerebral tumors.
* Uncountable seizures (clusters) or history of convulsive status epilepticus within the last five years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2003-11-24 (Actual); Primary Completion 2006-12-12 (Actual); Study Completion 2006-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (29):
- Hong Kong (3):
  - N01036 808, Hong Kong
  - N01036 842, Hong Kong
  - N01036 815, Kwun Tong
- Malaysia (3):
  - N01036 811, Kuala Lumpur
  - N01036 812, Kuala Lumpur
  - N01036 813, Kuala Lumpur
- Philippines (3):
  - N01036 830, Manila
  - N01036 831, Manila
  - N01036 829, Quezon
- Singapore (3):
  - N01036 804, Singapore
  - N01036 806, Singapore
  - N01036 807, Singapore
- Taiwan (12):
  - N01036 828, Changhua
  - N01036 827, Hualien City
  - N01036 825, Kaohsiung City
  - N01036 834, Kaohsiung City
  - N01036 835, Kaohsiung City
  - N01036 817, Taichung
  - N01036 823, Taichung
  - N01036 818, Tainan
  - N01036 819, Taipei
  - N01036 820, Taipei
  - N01036 821, Taipei
  - N01036 822, Taoyuan District
- Thailand (5):
  - N01036 809, Bangkok
  - N01036 840, Bangkok
  - N01036 841, Bangkok
  - N01036 839, Chiang Mai
  - N01036 810, Khon Kaen

REFERENCES:
- [Result] Kwan P, Lim SH, Chinvarun Y, Cabral-Lim L, Aziz ZA, Lo YK, Tonner F, Beh K, Edrich P; N01036 (SKATE II) Investigator Group. Efficacy and safety of levetiracetam as adjunctive therapy in adult patients with uncontrolled partial epilepsy: the Asia SKATE II Study. Epilepsy Behav. 2010 May;18(1-2):100-5. doi: 10.1016/j.yebeh.2010.03.016. Epub 2010 May 11. PMID 20462804
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in November 2003 and concluded in May 2006.
Pre-assignment Details: Participant Flow refers to the Intend-to-treat (ITT) Set.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 251
Completed | 218
Not Completed | 33
Not completed — Adverse Event | 14
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 2
Not completed — Intake of expired drug | 7
Not completed — Psychological trauma | 1
Not completed — Sponsor decision | 1
Not completed — Patient met exclusion criteria | 1
Not completed — Patient decision | 1
Not completed — Poor compliance, dilantin toxicity | 1
Not completed — Met exclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Intend-to-treat (ITT) Set.
Arm/Group | Levetiracetam
Number analyzed (Participants) | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 240
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.42 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Time Frame: From Baseline until Safety visit (two weeks after last dose; up to Week 18)
Measure: Number; unit: Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 251
Participants | 184

2. Secondary Outcome: Percentage Change From Historical Baseline in Partial (Type I) Seizure Frequency Per Week Over the Treatment Period
Description: Percentage change from baseline in partial (Type I) seizure frequency over the treatment period standardized to 1 week period.
  Type I Partial (focal, local) seizure frequency per week will be derived from the seizure count information recorded on the daily record card (e.g. date, number, type of epileptic seizures) and is defined as the number of seizures standardized to a 1 week period.
  A negative value in percent change from historical baseline indicates a decrease in partial (type I) seizure frequency from historical baseline.
Time Frame: Week 16, compared to Baseline
Population: Only subjects with partial (Type I) seizure frequency per week at baseline >= 0 and non-missing values on treatment period are included in the analysis.
  Subjects withdrawing from the study are included up to their early discontinuation visit.
Measure: Median (Inter-Quartile Range); unit: percentage changes
Arm/Group | Levetiracetam
Number analyzed (Participants) | 237
percentage changes | -48.34 [-89.96 to 6.19]

3. Secondary Outcome: Percentage Change From Historical Baseline in Total (Type I+II+III) Seizure Frequency Per Week Over the Treatment Period
Description: Percentage change from baseline in total (type I+II+III) seizure frequency over the treatment period standardized to 1 week period.
  Types I+II+III seizure frequency (Type I: Partial (focal, local), Type II: Generalized (convulsive or non-convulsive), Type III: Unclassified) per week will be derived from the seizure count information recorded on the daily record card (e.g. date, number, type of epileptic seizures) and is defined as the number of seizures standardized to a 1 week period.
  A negative value in percent change from historical baseline indicates a decrease in total (type I+II+III) seizure frequency from historical baseline.
Time Frame: Week 16, compared to Baseline
Population: Only subjects with total (Type I+II+III) seizure frequency per week at baseline >= 0 and non-missing values on treatment period are included in the analysis.
  Subjects withdrawing from the study are included up to their early discontinuation visit.
Measure: Median (Inter-Quartile Range); unit: percentage changes
Arm/Group | Levetiracetam
Number analyzed (Participants) | 243
percentage changes | -46.43 [-89.29 to 5.88]

4. Secondary Outcome: Percentage of Participants With 50% Response in Seizure Frequency Per Week at Week 16
Description: 50% response in seizure frequency per Week is defined as >=50% reduction in seizure frequency from Baseline.
  Types I+II+III seizure frequency (Type I: Partial (focal, local), Type II: Generalized (convulsive or non-convulsive), Type III: Unclassified) per week will be derived from the seizure count information recorded on the daily record card (e.g. date, number, type of epileptic seizures) and is defined as the number of seizures standardized to a 1 week period.
Time Frame: Week 16, compared to Baseline
Population: Only subjects with seizure frequency per week at baseline >= 0 and non-missing values on treatment period are taken into account for the responder rates. By convention, subjects with frequency per week at baseline equal to zero were considered as non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 243
percentage of participants
  Partial (Type I) seizures | 47.7
  Total (type I+II+III) seizures | 48.1

5. Secondary Outcome: Percentage of Participants With 100% Response in Seizure Frequency Per Week at Week 16
Description: 100% response in seizure frequency per Week is defined as 100% reduction in seizure frequency from Baseline.
  Types I+II+III seizure frequency (Type I: Partial (focal, local), Type II: Generalized (convulsive or non-convulsive), Type III: Unclassified) per week will be derived from the seizure count information recorded on the daily record card (e.g. date, number, type of epileptic seizures) and is defined as the number of seizures standardized to a 1 week period.
Time Frame: Week 16, compared to Baseline
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 243
percentage of participants
  Partial (Type I) seizures | 20.2
  Total (type I+II+III) seizures | 20.2

6. Secondary Outcome: Percentage of Patients With Categorized Change From Baseline in Severity of Illness
Description: The overall change in the severity of the subject's illness, compared to the subject's condition prior to the levetiracetam intake, was assessed by the Investigator using Investigator's Global Evaluation Scale (IGS). Categories are as following: Marked improvement; Moderate improvement; Slight improvement; No change; Slight worsening; Moderate worsening; Marked worsening.
Time Frame: Baseline, Week 16
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 251
percentage of participants
  Marked improvement | 34.1
  Moderate improvement | 25.3
  Slight improvement | 16.5
  No change | 17.7
  Slight worsening | 3.2
  Moderate worsening | 2.8
  Marked worsening | 0.4

7. Secondary Outcome: Retention Rate at Week 16
Description: Retention rate, defined as the number of subjects who were still on levetiracetam at Visit 5 (Week 16) or on the day before divided by the number of subjects in the ITT population.
Time Frame: Week 16
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 251
percentage of participants | 85.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 2 (week 2) until Safety Visit (up to 2 weeks after the last dose, up to 16 weeks).
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 15/251
Other Adverse Events (participants affected / at risk) | 136/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=251)
Bicytopenia (Blood and lymphatic system disorders) | 1
Adverse drug reaction (General disorders) | 1
Dengue fever (Infections and infestations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Convulsion (Nervous system disorders) | 4
Coordination abnormal (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Grand mal convulsion (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Anger (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam (N=251)
Nausea (Gastrointestinal disorders) | 14
Fatigue (General disorders) | 15
Dizziness (Nervous system disorders) | 36
Headache (Nervous system disorders) | 16
Sedation (Nervous system disorders) | 15
Somnolence (Nervous system disorders) | 75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days